CLINICAL TRIAL: NCT04510909
Title: COMMIT Depression Acceptability and Feasibility Trial
Brief Title: COMMIT Depression Trial Nepal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Possible (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, San Francisco (Other); Icahn School of Medicine at Mount Sinai, Department of Health Systems Design and Global Health (Unknown); Nyaya Health Nepal (Unknown); Ministry of Health and Population, Nepal (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: COMMITDNepal; 1R21MH116728-01A1 (NIH)
Record Dates: First submitted 2020-07-17; First posted 2020-08-12 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Depression
Keywords: low- and middle-income countries; mHealth; human-centered design and engineering; digital tools; Nepal; motivational interviewing; non-physician healthcare workers; community health workers; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot arm (Experimental): Mixed methods, acceptability and feasibility pilot of the COMMIT mHealth application
  Interventions: Other: COMMIT mHealth application

INTERVENTIONS:
Other: COMMIT mHealth application — The investigators will develop Community-based mHealth Motivational Interviewing Tool (COMMIT) using iterative design and testing with frequent, structured input from the key stakeholders: community health workers (CHWs), their supervisors and adult depression patients.The tool will be used by community CHWs in Dolakha, Nepal to: 1) obtain decision-support to deliver motivational interviewing (MI) for patients in their communities, and 2) capture consented audio recordings of client interactions for review and feedback by their supervisors, allowing CHWs to maintain MI skills beyond the initial training period.

SUMMARY:
Community health workers (CHWs) have successfully used Motivational Interviewing (MI) to improve treatment adherence (i.e. taking medications and attending clinic appointments) for patients with depression in the US and globally. Mobile health (mHealth) tools can address challenges in implementing MI by providing real-time support in the community and facilitating ongoing coaching and supervision for CHWs, as these two challenges currently impede CHWs' ability to use MI. The investigators will develop then test a new mHealth app, which can potentially be used in the US and abroad, to help CHWs receive decision-support for MI and capture consented audio recordings of patient interactions for review and feedback by facility-based nurses with MI expertise.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for patient population: a. Adult patients aged 18 or older; AND b. Must have with active diagnosis of moderate to severe depression (last PHQ-9 ≥10) in the electronic health record system at the research performance site in Nepal; AND c. Have poor adherence (did not refill medications 1 week past the expected date and/or missed a scheduled clinic visit by at least 2 weeks; AND d. Must reside in Dolakha, Nepal
2. Inclusion criteria for community health worker or a community health worker supervisor: a. community health workers and their supervisors currently employed by and working at the research performance site, serving communities in Dolakha; AND b. have received training in motivational interviewing and use of the COMMIT mobile application.

Exclusion Criteria:

1. Exclusion criteria for patient population: patients with bipolar disorder (their treatment will be different from standard antidepressants) and those with substance use or psychotic disorders (their motivational factors will be substantially different from those of other depressed patients).
2. Exclusion criteria for a community health worker or a community health worker supervisor: includes decision not to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Depression | 6 months
  Individual Patient Health Questionnaire-9 score, measured at baseline and endline, with greater than or equal to 10 as moderate to severe depression (min score=0; max scote=27 with higher score corresponding to poorer health status)
Medication refill percentage | 2 weeks
  Individual depression medication refill percentage over past 2 weeks (percentage of prescribed depression medication not refilled/picked up as measured by limited dataset extraction from electronic health record system; scale of 0-100%; minimum: 0%; maximum: 100%; higher scores correspond to medication refills completed 100% of the time).
Follow-up clinic attendance percentage | 2 weeks
  Individual attendance at follow-up visits measured as a percentage over past 2 weeks (percentage of indicated follow-up clinic visits that occurred as measured by limited dataset extraction from electronic health record system; scale of 0-100%; minimum: 0%; maximum: 100%; higher scores correspond to patients who attend follow-up visits at clinic 100% of the time).

SECONDARY OUTCOMES:
Application access and completion percentage | 6 months
  Frequency of community health worker accessing mobile application during study (number of times mobile application is accessed/data are entered and completed as a proportion of patients assigned for follow-up)
Patient encounter duration | 6 months
  Total amount of time spent using mobile application during patient encounter (amount of time spent in the application and at each prompt)
Application error/crash percentage | 6 months
  Frequency of mobile application displaying error messages or crashing while in use by community health workers during patient encounters (proportion of all patient encounters where an error message/application crashes occurs)

CONTACTS AND LOCATIONS:
Locations (1):
- Bayalpata Hospital, Sanfebagar-10, Achham/Province 7, Nepal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT04510909/ICF_000.pdf